CLINICAL TRIAL: NCT06755502
Title: Evaluation of Allium Sativum As Root Filling Material for Primary Molars Indicated for Non Vital Pulp Therapy: Randomized Clinical Trials
Brief Title: Garlic Oil As Root Filling Material in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennat Allah Ashraf Abd Elsabour Abd Elkareem, PhD degree student, Faculty of Dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 555
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Irreversible Pulpitis (toothache)
Keywords: RCT; garlic oil; natural remedies; primary molars; root canal filling material
MeSH Terms: conditions — Toothache | interventions — allyl sulfide; Calcium Hydroxide; iodoform; Ointments; Metapex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- garlic oil with zinc oxide group (Experimental)
  Interventions: Combination Product: Garlic oil
- metapex group (Active Comparator)
  Interventions: Drug: Calcium Hydroxide, Iodoform, paste

INTERVENTIONS:
Combination Product: Garlic oil — garlic oil mixed with zinc oxid powder, as root canal filling material
  Arms: garlic oil with zinc oxide group
Drug: Calcium Hydroxide, Iodoform, paste — Metapex as root canal filling materials
  Other Names: metapex
  Arms: metapex group

SUMMARY:
The goal of this study is to test garlic oil mixed with zinc oxide as a potential root canal filling material of primary molars in children aged from four to eight years.

the study hypothesized that garlic oil mixed with zinc oxide would be the same as the gold standard filling material (metapex).

The group receiving the garlic oil with zinc oxide as root canal filling material will be compared with other similar group receiving metapex as root canal filling material in terms of clinical and radio-graphic success, and working time.

DETAILED DESCRIPTION:
This study is a randomized clinical trial (RCT), that aims compare the clinical and radio-graphic success of garlic oil mixed with zinc oxide, used as root canal filling material in primary molars in children aged from four to eight years, with the conventional root filling material, which is metapex.

ELIGIBILITY:
Inclusion Criteria:

1. Primary second molars which are diagnosed with irreversible pulpitis, or pulp necrosis.
2. Presence of sinus tract.
3. Periapical bone swelling.
4. Continuous bleeding after amputation of the coronal pulp tissue.
5. No pulp tissue remains when the pulp chamber is accessed.
6. Pus discharges from the canal.
7. Radiographically, only primary molars with at least two-thirds of the root length.
8. Presence of inter-radicular or periapical radiolucency.

Exclusion Criteria:

1. A tooth with internal root resorption will not be included. 2. Excessive tooth mobility beyond healing. 3. Carious perforation in the pulpal flour. 4. A tooth with a pathological lesion extending to the successor's tooth germ. 5. Non-restorable primary molars.

-

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2026-10-08 (Estimated); Study Completion 2026-11-08 (Estimated)

PRIMARY OUTCOMES:
The clinical success rate | 3, 6,9,and 12 months
  The criteria of successful treatment, according to which the clinical evaluation will be done, will be "No abnormal mobility", "No sensitivity to percussion", and "No swelling"
Radio-graphic success | 6, and 12 month.
  For the radiographic success, the evaluation criteria will be "Preoperative pathological inter-radicular and/or periapical radiolucency started to resolve, or remained the same size", "No new postoperative pathological radiolucency developed", and "No pathological internal or external root resorption"

IPD SHARING:
Plan to Share IPD: Undecided